CLINICAL TRIAL: NCT00439504
Title: Double-Blind, Placebo-Controlled, Cross-Over Assessment of Intravenous Methamphetamine and Sublingual Lobeline Interactions
Brief Title: Ph1 Lobeline Interaction Study - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CPU-0012-1
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2007-02

CONDITIONS: Methamphetamine Dependence
MeSH Terms: interventions — Lobeline

INTERVENTIONS:
Drug: Lobeline

SUMMARY:
The purpose of this study is to determine if there are significant cardiovascular or other interactions between sublingual lobeline and intravenous methamphetamine.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 45 years of age
* Be in general good health with a history of methamphetamine (MA) abuse (but not dependence)
* If female and of child bearing potential, agrees to use birth control
* Be able to understand and provide written informed consent
* Have a body mass index between 18 and 30
* Have reported use of (MA) during the past three months without experiencing adverse consequence plus a life time MA or amphetamine use history of at least four occasions of use
* Have a negative drug test (barbiturates, benzodiazepines, amphetamines, opiates, cocaine, cannabinoids, ethanol) at screening and at the time of admission

Exclusion Criteria:

* Please contact site for details

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10

PRIMARY OUTCOMES:
Cardiovascular responses

SECONDARY OUTCOMES:
Subjective effects

CONTACTS AND LOCATIONS:
Overall Officials: Reese Jones, M.D., Principal Investigator — Langley Porter Psychiatric Institute
Locations (1):
- Langley Porter Psychiatric Institute, San Francisco, California, United States